CLINICAL TRIAL: NCT03676998
Title: Determinants of the Recovery of Diaphragm Dysfunction in Patients With Prolonged Mechanical Ventilation
Brief Title: Diaphragm Dysfunction During Prolonged Mechanical Ventilation
Acronym: DD-SRPR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: K171101J; 2017-A03091-52 (Other: ANSM)
Record Dates: First submitted 2018-08-10; First posted 2018-09-19 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Prolonged Mechanical Ventilation
Keywords: Prolonged weaning; Diaphragm dysfunction; Liberation from mechanical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Measurement of diaphragm function (Other): Patients will be followed up from admission to weaning with twice a week a diaphragm function multimodal evaluation (ultrasound, phrenic nerves stimulation technique)
  Interventions: Device: Measurement of diaphragm function

INTERVENTIONS:
Device: Measurement of diaphragm function — A bilateral magnetic stimulation induces a non voluntary diaphragm contraction and a drop in airway pressure that is measured.

SUMMARY:
The transition to unassisted breathing after invasive ventilation often proves challenging. Persistent ventilator dependence predisposes patients to nosocomial complications and death and increases the economic burden of critical illness. Ventilator-dependence results from an imbalance between the load and capacity of the respiratory muscle pump. Patients who fail a trial of spontaneous breathing commonly exhibit excess respiratory loads secondary to weaning-induced pulmonary edema, atelectasis or dynamic hyperinflation. At the same time, many ventilator-dependent patients exhibit striking loss of respiratory pump capacity due to diaphragm dysfunction which predisposes to prolonged ventilator dependence. Diaphragm dysfunction is common in ventilated patients. By prolonging ventilator dependence it may be an important contributor to the poor long-term clinical and functional outcomes of survivors of critical illness. While some main risk factors for diaphragm dysfunction have been already described (diaphragm disuse induced by mechanical ventilation, sepsis, initial severity upon admission), the determinants of recovery of diaphragm dysfunction are unknown, as well it has not been elucidated whether diaphragm function can simply improve after the acute phase of ICU admission. Therefore, the goal of this study is to investigate the time course evolution of diaphragm function in patients exposed to prolonged duration of mechanical ventilation (i.e. in a weaning center) and to determine which factors are associated with an improvement of the diaphragm function leading to a safe mechanical ventilation discontinuation.

DETAILED DESCRIPTION:
In this prospective study, all patients admitted to the weaning center of Pitié-Salpêtrière Hospital to undertake a weaning program will be closely followed up to assess twice a week their diaphragm function. Only one experimental group will be constituted. Diaphragm function will be assessed with both 1) the phrenic nerves stimulation technique and 2) diaphragm ultrasound (thickness, thickening fraction). The time course evolution of the diaphragm function over the stay will be investigated and all potential factors involved in the change in diaphragm function will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old;
* Admission in weaning center;
* Tracheostomy;
* Ventilator dependence as defined by clinical intolerance criteria under spontaneous - breathing (Boles et al. ERJ 2017);
* Oral consent

Exclusion Criteria:

* Contre indication to the phrenic nerves stimulation technique (pace maker);
* Impossible liberation from the ventilator (degenerative neuromuscular diseases; high level spinal injury);
* Pregnancy;
* No insurance coverage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2019-02-22 (Actual); Primary Completion 2024-10-22 (Estimated); Study Completion 2024-10-22 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients successfully liberated from the ventilator | After 7 days of spontaneous breathing
  Liberation from the ventilator will be defined after 7 days of spontaneous

SECONDARY OUTCOMES:
Diaphragm function | Twice a week, up to 4 weeks
  Diaphragm function will be defined as pressure generating capacity. In practice, it will be assessed by using the phrenic nerves stimulation technique. A bilateral magnetic stimulation of the phrenic nerves will be done and the drop in endotracheal pressure so generated will be measured (twitch pressure).
Partial liberation from mechanical ventilation | During hospitalization in Intensive Care Unit (ICU), up to 4 weeks
  Partial liberation from ventilation will be defined by spontaneous breathing without the ventilator through closed or opened tracheostomy collar for a period of time between 12 and 24 hours, the rest of the time, patients being under invasive or non invasive mechanical ventilation.
Proportion of patients with diaphragm dysfunction upon admission and upon discharge | From date of admission in ICU until the date of hospital discharge in ICU, assessed up to 4 weeks
  Proportion of patients with diaphragm dysfunction will be the ratio of patients with diaphragm dysfunction over the total number of patients enrolled in the study. Diaphragm dysfunction will be defined as a twitch pressure (endotracheal pressure generated by magnetic stimulation) below 11 cmH2O.

CONTACTS AND LOCATIONS:
Overall Officials: Martin DRES, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Pitié-Salpêtrière Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Virolle S, Duceau B, Morawiec E, Fosse Q, Nierat MC, Parfait M, Decavele M, Demoule A, Delemazure J, Dres M. Contribution and evolution of respiratory muscles function in weaning outcome of ventilator-dependent patients. Crit Care. 2024 Dec 18;28(1):421. doi: 10.1186/s13054-024-05172-y. PMID 39696360